CLINICAL TRIAL: NCT06510556
Title: Feasibility Study of the FARAFLEX Mapping and Pulsed Field Ablation (PFA) System in the Treatment of Persistent Atrial Fibrillation
Brief Title: Feasibility Study of the FARAFLEX Mapping and PFA System
Acronym: ELEVATE-PF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF306
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation; Paroxysmal AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Approximately 200 FARAFLEX treatment subjects will be enrolled and treated with the investigational FARAFLEX™ Mapping and PFA System. Approximately 50 commercial sub-study subjects will be enrolled and treated with a commercially approved PFA system per IFU and medical guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FARAFLEX Treatment group (Other): 200 subjects scheduled to undergo endocardial mapping and ablation in the treatment of persistent atrial fibrillation or paroxysmal atrial fibrillation with FARAFLEX mapping PFA catheter and other BSC devices.
  Interventions: Device: FARAFLEX Ablation Treatment
- Commercial sub-study group (Other): Approximately 50 subjects meeting study eligibility requirements will be enrolled in a commercial sub-study at a subset of centers and will undergo endocardial mapping and ablation in the treatment of persistent atrial fibrillation or paroxysmal atrial fibrillation with a commercially approved PFA systems.
  Interventions: Device: Commercial Sub-study Treatment

INTERVENTIONS:
Device: FARAFLEX Ablation Treatment — Subjects scheduled to undergo endocardial mapping and ablation therapy in the treatment of persistent atrial fibrillation or paroxysmal atrial fibrillation. Using the investigational Boston Scientific FARAFLEX Mapping and Pulse Field Ablation (PFA) System, ablation of the pulmonary veins will be performed; ablation of the left atrial posterior wall, mitral isthmus (MI), LA roof line and/or cavo-tricuspid isthmus (CTI) is at the discretion of the investigator.
  Arms: FARAFLEX Treatment group
Device: Commercial Sub-study Treatment — Subjects scheduled to undergo endocardial mapping and ablation therapy in the treatment of persistent atrial fibrillation or paroxysmal atrial fibrillation. Using a commercially available PFA system, ablation of the pulmonary veins will be performed; ablation of the left atrial posterior wall, mitral isthmus (MI), LA roof line and/or cavo-tricuspid isthmus (CTI) is at the discretion of the investigator, per the selected catheter's IFU and in accordance with the guidelines.
  Arms: Commercial sub-study group

SUMMARY:
The objective of this feasibility study is to evaluate the safety and effectiveness of the FARAFLEX mapping and pulsed field ablation (PFA) catheter, a novel catheter in treating persistent atrial fibrillation (PersAF) or symptomatic Paroxysmal Atrial Fibrillation (PAF).

DETAILED DESCRIPTION:
The objective of this study is to obtain First-in-Human (FIH) experience with the FARAFLEX mapping and PFA catheter in the treatment of persistent Atrial Fibrillation (persAF) or Paroxysmal Atrial Fibrillation (PAF).

Subjects with symptomatic Persistent Atrial Fibrillation or symptomatic Paroxysmal Atrial Fibrillation will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age, or older if required by local law
2. Symptomatic, documented, Persistent AF or Paroxysmal AF
3. Willing and capable of providing informed consent
4. Willing and capable of participating in all follow-up assessments and testing associated with this clinical investigation at an approved clinical investigational center

Exclusion Criteria:

1. Atrial exclusions - Any of the following atrial conditions:

   * Left atrial anteroposterior diameter ≥ 5.5 cm, or if LA diameter not available, non indexed volume >100 ml (by MRI, CT or TTE report or physician note)
   * Any prior atrial endocardial, epicardial or surgical ablation procedure for atrial arrhythmia other than ablation for right sided SVT
   * Current atrial myxoma
   * Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   * Current left atrial thrombus
2. Cardiovascular exclusions - Any of the following CV conditions:

   * History of sustained ventricular tachycardia or any ventricular fibrillation AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   * Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, interatrial baffle, closure device, patch, or patent foramen ovale occluder, LA appendage closure, device or occlusion
   * Valvular disease that is symptomatic or is the cause of heart failure.
   * Hypertrophic cardiomyopathy
   * Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty
   * Known inability to obtain vascular access or other contraindication to femoral access
   * Rheumatic heart disease
   * Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
   * Known allergic drug reaction to nitroglycerin1
   * Known severe non-revascularizable coronary disease
   * Pre-existing right coronary artery stent and left circumflex artery
3. Any of the following conditions at baseline:

   * Heart failure associated with NYHA Class IV
   * LVEF < 40%
   * Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two (2) BP measurements at baseline assessment
   * Severe right ventricular dysfunction with documented echocardiography and/or hemodynamic data.
4. Any of the following events within 90 Days of the Consent Date:

   * Myocardial infarction (MI), unstable or Prinzmetal angina or coronary intervention
   * Any cardiac surgery
   * Heart failure hospitalization
   * Pericarditis or symptomatic pericardial effusion
   * Gastrointestinal bleeding
   * Stroke, TIA, or intracranial bleeding
   * Any non-neurologic thromboembolic event
   * Carotid stenting or endarterectomy
5. Known coagulopathy disorder (e.g. von Willibrand's disease, hemophilia)
6. Contraindication to, or unwillingness to use, systemic anticoagulation, or acceptable alternatives, pre-, intra- and post-procedure to achieve adequate anticoagulation.
7. Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
8. Any of the following health conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:

   * Body Mass Index (BMI) > 42.0
   * Solid organ or hematologic transplant, or currently being evaluated for a transplant
   * Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
   * Severe lung disease, severe pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   * Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   * Active malignancy at enrollment (other than squamous cell carcinoma)
   * Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   * Active systemic infection
   * Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour)
   * Required use of phosphodiesterase inhibitors within 24 hours of the ablation procedure

10. Predicted life expectancy less than one (1) year 11. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility 12. Any of the following congenital conditions:

* Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
* History of known congenital methemoglobinemia
* History of known G6PD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Device or procedure-related Composite Serious Adverse Events (CSAEs) | Ablation Procedure (Day 0) - Day 7; Day 0- Day 30; Day 0- Day 360
  the incidence of device or procedure-related Composite Serious Adverse Events (CSAEs) following the Index Procedure will be evaluated. Safety analyses will be reported by AF type (Paroxysmal vs. Persistent) and treatment group (FARAFLEX vs. Commercial catheter).
Acute Procedural Success | At the end of the ablation procedure
  The proportion of subjects that achieve Acute Procedural Success (APS) defined as the percutaneous endocardial creation of a complete, electrically isolating set of lesions around the ostia of the pulmonary veins (PV) and the posterior wall (PW) during the Index Procedure, as clinically assessed by entrance and/or exit block. Effectiveness analyses will be reported by AF type (Paroxysmal vs. Persistent) and treatment group (FARAFLEX vs. Commercial catheter).

CONTACTS AND LOCATIONS:
Locations (3):
- Klinicki bolnicki centar Split, Split, Croatia
- Nemocnice Na Homolce Hospital, Prague, Czechia
- Fondazione PTV - Policlinico Tor Vergata, Roma, Italy